CLINICAL TRIAL: NCT02991495
Title: A Randomized, Blinded Non-inferiority Trial on the Immunogenicity and Safety of Fractional Doses of Yellow Fever Vaccines in Kenya and Uganda
Brief Title: Immunogenicity and Safety of Fractional Doses of Yellow Fever Vaccines (YEFE)
Acronym: YEFE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Epicentre (Other)
Collaborators: Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: YEFE_2017
Record Dates: First submitted 2016-12-07; First posted 2016-12-13 (Estimated); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Yellow Fever
Keywords: Epidemic response
MeSH Terms: conditions — Yellow Fever | interventions — Yellow Fever Vaccine; Seroconversion

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Stamaril, Sanofi Pasteur: Standard dose (Active Comparator): Subcutaneous administration of 1 dose of a standard yellow fever vaccine
  Interventions: Biological: Stamaril, Sanofi Pasteur
- Stamaril, Sanofi Pasteur: Fractional dose (Experimental): Subcutaneous administration of 1/5th of a standard dose of yellow fever vaccine
  Interventions: Biological: Stamaril, Sanofi Pasteur
- Yellow fever vaccine, Bio-Manguinhos: Standard dose (Active Comparator): Subcutaneous administration of 1 dose of a standard yellow fever vaccine
  Interventions: Biological: Yellow fever vaccine, Bio-Manguinhos
- Yellow fever vaccine, Bio-Manguinhos: Fractional dose (Experimental): Subcutaneous administration of 1/5th of a standard dose of yellow fever vaccine
  Interventions: Biological: Yellow fever vaccine, Bio-Manguinhos
- Yellow fever vaccine, Institut Pasteur: Standard dose (Active Comparator): Subcutaneous administration of 1 dose of a standard yellow fever vaccine
  Interventions: Biological: Yellow fever vaccine, Institut Pasteur
- Yellow fever vaccine, Institut Pasteur: Fractional dose (Experimental): Subcutaneous administration of 1/5th of a standard dose of yellow fever vaccine
  Interventions: Biological: Yellow fever vaccine, Institut Pasteur
- Yellow fever vaccine, Chumakov Institute: Standard dose (Active Comparator): Subcutaneous administration of 1 dose of a standard yellow fever vaccine
  Interventions: Biological: Yellow fever vaccine, Chumakov Institute
- Yellow fever vaccine, Chumakov Institute: Fractional dose (Experimental): Subcutaneous administration of 1/5th of a standard dose of yellow fever vaccine
  Interventions: Biological: Yellow fever vaccine, Chumakov Institute
- YF, Chumakov Institute: Standard dose in Children (Active Comparator): Subcutaneous administration of 1 dose of the yellow fever vaccine
  Interventions: Biological: Yellow fever vaccine, Chumakov Institute
- YF, Chumakov Institute: Fractional dose in Children (Experimental): Subcutaneous administration of 1/5th of a standard dose of yellow fever vaccine
  Interventions: Biological: Yellow fever vaccine, Chumakov Institute
- YF, Chumakov Institute: Standard dose in HIV+ adults (Active Comparator): Subcutaneous administration of 1 dose of the yellow fever vaccine
  Interventions: Biological: Yellow fever vaccine, Chumakov Institute
- YF, Chumakov Institute: Fractional dose in HIV+ adults (Experimental): Subcutaneous administration of 1/5th of a standard dose of yellow fever vaccine
  Interventions: Biological: Yellow fever vaccine, Chumakov Institute

INTERVENTIONS:
Biological: Stamaril, Sanofi Pasteur — 1. Full dose
  2. Fractional dose: one fifth (1/5)
  Arms: Stamaril, Sanofi Pasteur: Fractional dose; Stamaril, Sanofi Pasteur: Standard dose
Biological: Yellow fever vaccine, Bio-Manguinhos — 1. Full dose
  2. Fractional dose: one fifth (1/5)
  Arms: Yellow fever vaccine, Bio-Manguinhos: Fractional dose; Yellow fever vaccine, Bio-Manguinhos: Standard dose
Biological: Yellow fever vaccine, Institut Pasteur — 1. Full dose
  2. Fractional dose: one fifth (1/5)
  Arms: Yellow fever vaccine, Institut Pasteur: Fractional dose; Yellow fever vaccine, Institut Pasteur: Standard dose
Biological: Yellow fever vaccine, Chumakov Institute — 1. Full dose
  2. Fractional dose: one fifth (1/5)
  Arms: Yellow fever vaccine, Chumakov Institute: Fractional dose; Yellow fever vaccine, Chumakov Institute: Standard dose
Biological: Yellow fever vaccine, Chumakov Institute — 1. Full dose
  2. Fractional dose: one fifth (1/5)
  Other Names: Children sub-study
  Arms: YF, Chumakov Institute: Fractional dose in Children; YF, Chumakov Institute: Standard dose in Children
Biological: Yellow fever vaccine, Chumakov Institute — 1. Full dose
  2. Fractional dose: one fifth (1/5)
  Other Names: HIV + adults
  Arms: YF, Chumakov Institute: Fractional dose in HIV+ adults; YF, Chumakov Institute: Standard dose in HIV+ adults

SUMMARY:
In July 2016, the demand for yellow fever vaccines in response to the large urban outbreaks occurring concurrently and the risk of further spread through the African continent and even to Asia, was larger than the available supply. In this situation, the World Health Organization (WHO) developed recommendations for the use of fractional-dose of yellow fever vaccine as a dose-sparing strategy. These recommendations were based on limited number of clinical trials and additional studies should assess the applicability of the fractional dose to all WHO-prequalified vaccines, the persistence of neutralizing antibodies and the performance of the fractional dose in young children and populations in Africa including those with HIV.

This study aims to respond to some of the research questions that would allow broadening the recommendations on the use of fractional doses of yellow fever vaccine in emergency situations. The study will be conducted in Uganda and Kenya and the main objective is to assess the non-inferiority is seroconversion 28 days after vaccination of a fractional dose compared to full dose for each WHO-prequalified manufacturer. As secondary objectives the study will assess seroprotection 10 days and 1 year after vaccination, to assess rapidity and persistence of protective antibody levels; describe the geometric mean titre and the change in neutralizing antibody on Day 28 days after vaccination with fractional and full doses; and assess the occurrence of adverse events and serious adverse events (SAE) during 28 days after administration of fractional and full doses.

The study consists of a randomized non-inferiority trial. The study aims to start in April 2017 in the two sites and aims to recruit 960 adults. Results for the main outcome will be reviewed by the study Data and Safety Monitoring Board and one vaccine will be selected for the studies in children and HIV positive adults.

DETAILED DESCRIPTION:
Yellow fever (YF) is a mosquito-borne viral disease that is endemic in 34 countries in the African region and 14 in South America. YF virus infection can be asymptomatic or cause a wide spectrum of disease, from mild symptoms to severe, potentially lethal illness with jaundice, renal failure and haemorrhage. The vast majority of reported cases and deaths occur in sub-Saharan Africa where yellow fever is a major health problem occurring in epidemic patterns. There is no specific treatment for yellow fever infection. However, YF vaccine is shown to be very effective for outbreak control as well as for the prevention of outbreaks. YF vaccination confers protection in most vaccinated individuals and this is considered to be life-long.

In 2016, YF outbreaks occurred in Africa (Angola, Democratic Republic of Congo (DRC) and Uganda) as well as in South America (Brazil, Colombia and Peru). Factors such increased urbanization in poor areas without proper water and sanitation systems and population movements, have the potential to contribute to increasing incidence of yellow fever and large epidemics. In July 2016, the demand for yellow fever vaccines in response to the large urban outbreaks occurring concurrently and the risk of further spread through the African continent and even to Asia, was larger than the available supply. In this situation, the World Health Organization (WHO) developed recommendations for the use of fractional-dose of yellow fever vaccine as a dose-sparing strategy. This strategy consisted on delivering 1/5th of the conventional dose and was used to vaccinate over 7 million people in Kinshasa, the capital city of DRC.

The evidence to recommend the use of fractional dosing was based on a limited number of clinical studies. However this was considered sufficient to provide emergency recommendations. In order to broaden and also possibly simplify WHO recommendations of fractional dose use in case of need for emergency campaigns, additional data is needed to respond to the important data gaps. These include the applicability of the fractional dose to all WHO-prequalified vaccines, the persistence of neutralizing antibodies and the performance of the fractional dose in young children and populations in Africa including those with HIV. Following these data gaps, WHO called for research to be conducted.

This study aims to respond to some of the research questions that would allow to broaden the recommendations on the use of fractional doses of yellow fever vaccine in emergency situations. The study will be conducted in Uganda and Kenya and the main objective is to assess the non-inferiority is seroconversion 28 days after vaccination of a fractional dose compared to full dose for each manufacturer. As secondary objectives the study will assess seroprotection 10 days and 1 year after vaccination, to assess rapidity and persistence of protective antibody levels; describe the geometric mean titre and the change in neutralizing antibody on Day 28 after vaccination with fractional and full doses; and assess the occurrence of adverse events and serious adverse events (SAE) during 28 days after administration of fractional and full doses. The study aims to recruit 960 adults (480 in Mbarara, Uganda, and 480 in Kilifi, Kenya). Results for the main outcome will be reviewed by the study Data and Safety Monitoring Board (DSMB) and if results are considered satisfactory, the study will continue with the recruitment of 420 children in Uganda and 250 HIV infected adults in Kenya, to assess non-inferiority of one of the WHO prequalified vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Adults population: 18 to 60 years of age
* Children population: 9 to 59 months of age
* For HIV positive population: HIV positive on serological testing
* If HIV infection, CD4 T-cell counts ≥200 cells/mm³ for adults or CD4 percentage >25% for children
* Providing informed consent to participate in the study

Exclusion Criteria:

* Contraindications to yellow fever vaccination:
* History of yellow fever vaccination
* Previous yellow fever infection
* Requiring yellow fever vaccination for travelling purposes
* Pregnancy (as determined by a urine test on the proposed day of vaccination) and lactating women
* Refusal to participate in the study
* Planning to move out of the study area before the end of the study follow-up

Ages: 9 Months to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1630 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Seroconversion by PRNT50 (Plaque Reduction Neutralization Test 50 value) | 28 days post-vaccination
  Plaque reduction neutralization test will be used to quantify the titer of neutralising antibody for the virus

SECONDARY OUTCOMES:
Assessment of protection by PRNT50 (Plaque Reduction Neutralization Test 50 value) | 10 days post-vaccination
  Plaque reduction neutralization test will be used to quantify the titer of neutralising antibody for the virus
Duration of immunity | 1 year post-vaccination
  Assessment of duration of immunity at 1 year after vaccination
Assessment of adverse events and serious adverse events | 28 days post-vaccination

CONTACTS AND LOCATIONS:
Locations (2):
- KEMRI, Kilifi, Kenya
- Epicentre, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Juan-Giner A, Namulwana ML, Kimathi D, Grantz KH, Fall G, Dia M, Bob NS, Sall AA, Nerima C, Sahani MK, Mulogo EM, Ampeire I, Hombach J, Nanjebe D, Mwanga-Amumpaire J, Cummings DAT, Bejon P, Warimwe GM, Grais RF. Immunogenicity and safety of fractional doses of 17D-213 yellow fever vaccine in children (YEFE): a randomised, double-blind, non-inferiority substudy of a phase 4 trial. Lancet Infect Dis. 2023 Aug;23(8):965-973. doi: 10.1016/S1473-3099(23)00131-7. Epub 2023 Apr 28. PMID 37127047
- [Derived] Kimathi D, Juan-Giner A, Orindi B, Grantz KH, Bob NS, Cheruiyot S, Hamaluba M, Kamau N, Fall G, Dia M, Mosobo M, Moki F, Kiogora K, Chirro O, Thiong'o A, Mwendwa J, Guantai A, Karanja HK, Gitonga J, Mugo D, Ramko K, Faye O, Sanders EJ, Grais RF, Bejon P, Warimwe GM. Immunogenicity and safety of fractional doses of 17D-213 yellow fever vaccine in HIV-infected people in Kenya (YEFE): a randomised, double-blind, non-inferiority substudy of a phase 4 trial. Lancet Infect Dis. 2023 Aug;23(8):974-982. doi: 10.1016/S1473-3099(23)00114-7. Epub 2023 Apr 28. PMID 37127045
- [Derived] Juan-Giner A, Kimathi D, Grantz KH, Hamaluba M, Kazooba P, Njuguna P, Fall G, Dia M, Bob NS, Monath TP, Barrett AD, Hombach J, Mulogo EM, Ampeire I, Karanja HK, Nyehangane D, Mwanga-Amumpaire J, Cummings DAT, Bejon P, Warimwe GM, Grais RF. Immunogenicity and safety of fractional doses of yellow fever vaccines: a randomised, double-blind, non-inferiority trial. Lancet. 2021 Jan 9;397(10269):119-127. doi: 10.1016/S0140-6736(20)32520-4. PMID 33422245
- [Derived] Kimathi D, Juan A, Bejon P, Grais RF, Warimwe GM; YEFE and NIFTY vaccine trials teams. Randomized, double-blinded, controlled non-inferiority trials evaluating the immunogenicity and safety of fractional doses of Yellow Fever vaccines in Kenya and Uganda. Wellcome Open Res. 2019 Nov 20;4:182. doi: 10.12688/wellcomeopenres.15579.1. eCollection 2019. PMID 31984244